CLINICAL TRIAL: NCT05694013
Title: Interventional Platform Study Investigating the Impact of Digital Health Solutions on Health Outcomes and Health-Care Resource Utilization in Participants Receiving Systemic Treatment in Clinical Practice
Brief Title: Clinical Impact and Utility of Digital Health Solutions in Participants Receiving Systemic Treatment in Clinical Practice
Acronym: ORIGAMA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study terminated by sponsor.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO42720
Record Dates: First submitted 2022-12-20; First posted 2023-01-23 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Cancer
Keywords: Remote Patient Monitoring, Digital Patient Monitoring, Symptom Monitoring, Digital Health
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A - Arm 1 (Experimental): Participants with metastatic non-small cell lung carcinoma (mNSCLC), extensive-stage small-cell lung carcinoma (ES-SCLC), and advanced or unresectable hepatocellular carcinoma (HCC) and who are prescribed an anticancer regimen including intravenous (IV) atezolizumab will use the Roche Digital Patient Monitoring (DPM) Module along with local standard of care (SOC) support.
  Interventions: Device: Roche DPM Module; Other: Local SOC support
- Cohort A - Arm 2 (Experimental): Participants with mNSCLC, ES-SCLC, and HCC who are prescribed an anticancer regimen including IV atezolizumab will receive local SOC support.
  Interventions: Other: Local SOC support
- Cohort B (Experimental): Participants with resected Stage IIB-IIIB NSCLC will use the Roche DPM Module along with subcutaneous (SC) atezolizumab in both the hospital and flexcare (home) setting.
  Interventions: Device: Roche DPM Module; Drug: Atezolizumab SC

INTERVENTIONS:
Device: Roche DPM Module — Participants will be trained in the use of the Roche DPM Module, which they will use alongside local SOC support
  Arms: Cohort A - Arm 1; Cohort B
Drug: Atezolizumab SC — Participants will receive atezolizumab SC for 16 cycles (cycle length = 21 days)
  Arms: Cohort B
Other: Local SOC support — Participants will receive local SOC support
  Arms: Cohort A - Arm 1; Cohort A - Arm 2

SUMMARY:
This study will evaluate the clinical impact and utility of digital health solutions (DHS) on health outcomes and health-care resource utilization in people receiving systemic anti-cancer treatment (approved or non-approved) in clinical practice.

ELIGIBILITY:
Inclusion Criteria: All Participants

* Email address, access to an internet-capable device (smartphone, tablet, or PC), and access to an internet connection

Inclusion Criteria: Cohort A

* Histologically confirmed diagnosis for mNSCLC, ES-SCLC, or HCC (Child Pugh A)
* Systemic therapy naive
* Prescribed an atezolizumab IV regimen
* Easter Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2

Inclusion Criteria: Cohort B

* Complete resection of a histologically or cytologically confirmed Stage IIB-IIIB (T3-N2) NSCLC
* PD-L1 positive
* Have completed adjuvant chemotherapy at least 4 weeks and up to 12 weeks prior to randomization and must be adequately recovered from chemotherapy treatment
* ECOG Performance Status of 0 or 1
* Adequate hematologic and end-organ function
* For participants receiving therapeutic anticoagulation: stable anticoagulant regimen
* Negative for hepatitis B virus (HBV) or hepatitis C virus (HCV)

Exclusion Criteria: All Participants

* Any physical or cognitive condition that would prevent the participant from using the DHS
* Participants not proficient with any of the available DHS language translations or with psychiatric/neurologic disorders or any condition that may impact the participant's ability to use the DPM solution
* Currently participating in another interventional trial
* History of malignancy within 5 years prior to initiation of study treatment, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death

Exclusion Criteria: Cohort A

* Concomitant anti-cancer therapy at the time of starting atezolizumab (IV) regimen on the index date which is not part of a locally approved combination therapy with atezolizumab
* Participants not receiving atezolizumab, but an atezolizumab biosimilar or non-comparable biologic
* Participants currently using another DPM or ePRO solution for symptom management and/or reporting

Exclusion Criteria: Cohort B

* Participants known to have a sensitizing mutation in the EGFR gene or an ALK fusion oncogene
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* History of leptomeningeal disease
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active tuberculosis
* Significant cardiovascular disease
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact participant safety
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* Prior allogeneic stem cell or solid organ transplantation
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Current treatment with anti-viral therapy for HBV
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2) within 4 weeks or 5 drug elimination half-lives (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-α [TNF-α] agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Pregnancy or breastfeeding
* Known allergy or hypersensitivity to hyaluronidase, bee or vespid venom, or any other ingredient in the formulation of rHuPH20
* Pathology (e.g., lower extremity edema, cellulitis, lymphatic disorder or prior surgery, preexisting pain syndrome, previous lymph node dissection, etc.) that could interfere with any protocol-specified outcome assessment
* Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 2 weeks prior to randomization
* Participants currently using another DPM or ePRO solution for symptom management and/or reporting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-LaRoche
Locations (14):
- Australia (4):
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Monash Medical Centre Clayton, Clayton, Victoria
  - Latrobe Regional Hospital, Traralgon, Victoria
- Austria (2):
  - Lkh-Univ. Klinikum Graz, Graz
  - Klinikum Klagenfurt am Wörtersee, Klagenfurt
- Germany (3):
  - Hämato-Onkologische Schwerpunktpraxis am Klinikum Aschaffenburg, Aschaffenburg
  - MVZ für Hämatologie, Onkologie, Strahlentherapie und Palliativmedizin -, Stade
  - Helios Klinik Wuppertal, Wuppertal
- Spain (3):
  - Hospital del Mar, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico, Jaén
- Switzerland (2):
  - Hôpital Universitaire de Genève (HUG), Geneva
  - CHUV, Lausanne

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Iivanainen S, Baird AM, Balas B, Bustillos A, Castro Sanchez AY, Eicher M, Golding S, Mueller-Ohldach M, Reig M, Welslau M, Ammann J. Assessing the impact of digital patient monitoring on health outcomes and healthcare resource usage in addition to the feasibility of its combination with at-home treatment, in participants receiving systemic anticancer treatment in clinical practice: protocol for an interventional, open-label, multicountry platform study (ORIGAMA). BMJ Open. 2023 Apr 19;13(4):e063242. doi: 10.1136/bmjopen-2022-063242. PMID 37076159

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with extensive- stage small-cell lung carcinoma (ES-SCLC) or hepatocellular carcinoma (HCC) or non-small cell lung carcinoma (NSCLC) that are prescribed a locally-approved anti-cancer regimen containing IV atezolizumab.
Groups:
- Atezolizumab Regimen: Participants with metastatic non-small cell lung carcinoma (mNSCLC) or extensive-stage small-cell lung carcinoma (ES-SCLC) or advanced or unresectable hepatocellular carcinoma (HCC) and who were prescribed an anticancer regimen including intravenous (IV) atezolizumab received local standard of care (SOC) support.
- Atezolizumab Regimen + DPM: Participants with mNSCLC or ES-SCLC or HCC who were prescribed an anticancer regimen including IV atezolizumab used the Roche Digital Patient Monitoring (DPM) Module along with local SOC support.
Period: Overall Study
Arm/Group | Atezolizumab Regimen | Atezolizumab Regimen + DPM
Started | 25 | 24
Completed | 3 | 3
Not Completed | 22 | 21
Not completed — Death | 6 | 2
Not completed — Participant Decision | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Progressive Disease | 0 | 1
Not completed — Study Terminated by Sponsor | 12 | 17
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab Regimen | Atezolizumab Regimen + DPM | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.1 (7.3) | 62.0 (8.5) | 65.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 18 | 15 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 19 | 12 | 31
  Unknown or Not Reported | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 23 | 23 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Global Health Status Score/Quality of Life Score (GHS/QoL) From the European Organisation for Research and Treatment of Cancer (EORTC) Item Library 6 (IL6) GHS/QoL
Description: The European Organisation for Research and Treatment of Cancer quality of life core questionnaire (EORTC QLQ-C30) consists of 30 questions that assess five aspects of patient functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), global health status (GHS) and quality of life (QoL), and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. The EORTC item library 6 (IL6) GHS/QoL consists of only the GHS and QoL items from the EORTC QLQ-C30. The raw score is calculated as the value of both answers, scored on a 7-point scale that ranges from 1 ("very poor") to 7 ("excellent"), then a linear transformation is applied to produce a score between 0-100. Higher scores indicate a higher QoL.
Time Frame: Baseline, Cycle 3 Day 1, Cycle 5 Day 1, Cycle 7 Day 1, Cycle 9 Day 1, Long Term Follow Up/Week 28 (cycle length = 21 days)
Population: The ITT population included all randomized participants.
Measure: Median (Full Range); unit: Units on a scale
Groups:
- Atezolizumab Regimen: Participants with metastatic non-small cell lung carcinoma (mNSCLC), extensive-stage small-cell lung carcinoma (ES-SCLC), and advanced or unresectable hepatocellular carcinoma (HCC) and who were prescribed an anticancer regimen including intravenous (IV) atezolizumab received local standard of care (SOC) support.
- Atezolizumab Regimen + DPM: Participants with mNSCLC, ES-SCLC, and HCC who were prescribed an anticancer regimen including IV atezolizumab used the Roche Digital Patient Monitoring (DPM) Module along with local SOC support.
Arm/Group | Atezolizumab Regimen | Atezolizumab Regimen + DPM
Number analyzed (Participants) | 25 | 24
Units on a scale
  Baseline: number analyzed (Participants) | 23 | 18
  Baseline | 66.67 [16.7 to 100.0] | 66.67 [33.3 to 100.0]
  Cycle 3 Day 1: number analyzed (Participants) | 15 | 20
  Cycle 3 Day 1 | 66.67 [16.7 to 100.0] | 58.33 [0.0 to 100.0]
  Cycle 5 Day 1: number analyzed (Participants) | 14 | 14
  Cycle 5 Day 1 | 62.50 [50.0 to 100.0] | 70.83 [41.7 to 100.0]
  Cycle 7 Day 1: number analyzed (Participants) | 10 | 8
  Cycle 7 Day 1 | 66.67 [25.0 to 100.0] | 83.33 [41.7 to 100.0]
  Cycle 9 Day 1: number analyzed (Participants) | 6 | 8
  Cycle 9 Day 1 | 62.50 [50.0 to 100.0] | 83.33 [66.7 to 91.7]
  Long Term Follow Up (Week 28): number analyzed (Participants) | 2 | 0
  Long Term Follow Up (Week 28) | 75.00 [50.0 to 100.0] |

2. Secondary Outcome: Change From Baseline in the EuroQol 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) Visual Analogue Scale (VAS) Instrument
Description: The EQ-5D-5L is used to calculate a health status utility score for use in health economic analyses. The questionnaire is designed to capture the participant's current health status. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, as well as a VAS that measures health state. The score range is 0-100, with higher scores indicating better outcomes.
Time Frame: as for outcome 1
Population: The ITT population consisted of all randomized participants.
Measure: Median (Full Range); unit: Units on a scale
Groups:
- Atezolizumab Regimen + DPM: Participants with mNSCLC, ES-SCLC, and HCC who are prescribed an anticancer regimen including IV atezolizumab will receive local SOC support.
Arm/Group | Atezolizumab Regimen | Atezolizumab Regimen + DPM
Number analyzed (Participants) | 25 | 24
Units on a scale
  Baseline: number analyzed (Participants) | 23 | 18
  Baseline | 71.00 [0.0 to 100.0] | 83.50 [31.0 to 100.0]
  Cycle 3 Day 1: number analyzed (Participants) | 15 | 21
  Cycle 3 Day 1 | 65.00 [2.0 to 96.0] | 59.00 [20.0 to 100.0]
  Cycle 5 Day 1: number analyzed (Participants) | 14 | 15
  Cycle 5 Day 1 | 78.00 [3.0 to 100.0] | 85.00 [37.0 to 100.0]
  Cycle 7 Day 1: number analyzed (Participants) | 10 | 10
  Cycle 7 Day 1 | 67.50 [32.0 to 99.0] | 65.00 [21.0 to 97.0]
  Cycle 9 Day 1: number analyzed (Participants) | 6 | 8
  Cycle 9 Day 1 | 67.50 [59.0 to 100.0] | 90.00 [49.0 to 94.0]
  Long Term Follow Up (Week 28): number analyzed (Participants) | 2 | 0
  Long Term Follow Up (Week 28) | 70.00 [40.0 to 100.0] |

3. Secondary Outcome: Change From Baseline in Mean Symptom Severity Score From the MDASI Core Items
Description: The MDASI assesses symptom severity and symptom interference with different aspects of a patient's life as rated by the patient. For 6 items (pertaining to patient's general activity, walking, work, mood, relations with other people and enjoyment of life), patients rate how the symptoms interfere with different aspects of their life in the last 7 days. The MDASI items are rated from 0-10, with 0 indicating that the symptom is either not present or does not interfere with the patient's activities and 10 indicating that the symptom is "as bad as you can imagine" or "interfered completely" with the patient's life.
Time Frame: as for outcome 1
Population: The ITT population consisted of all randomized participants.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Atezolizumab Regimen | Atezolizumab Regimen + DPM
Number analyzed (Participants) | 25 | 24
Units on a scale
  Baseline: number analyzed (Participants) | 25 | 20
  Baseline | 3.33 [0.0 to 9.8] | 3.08 [0.0 to 9.5]
  Cycle 3 Day 1: number analyzed (Participants) | 17 | 21
  Cycle 3 Day 1 | 2.67 [0.0 to 9.2] | 3.00 [0.0 to 8.0]
  Cycle 5 Day 1: number analyzed (Participants) | 15 | 15
  Cycle 5 Day 1 | 3.00 [0.0 to 9.0] | 2.33 [0.0 to 7.0]
  Cycle 7 Day 1: number analyzed (Participants) | 11 | 11
  Cycle 7 Day 1 | 1.50 [0.0 to 7.2] | 3.17 [0.0 to 5.8]
  Cycle 9 Day 1: number analyzed (Participants) | 6 | 11
  Cycle 9 Day 1 | 1.67 [0.0 to 5.0] | 1.17 [0.0 to 6.3]
  Long Term Follow Up (Week 28): number analyzed (Participants) | 2 | 0
  Long Term Follow Up (Week 28) | 3.42 [0.0 to 6.8] |

4. Secondary Outcome: Number of Cumulative Days Hospitalized Due to SAEs
Time Frame: Up to approximately 16 months
Population: The ITT population consisted of all randomized participants.
Measure: Median (Full Range); unit: Days
Arm/Group | Atezolizumab Regimen | Atezolizumab Regimen + DPM
Number analyzed (Participants) | 7 | 12
Days | 11.0 [4 to 30] | 4.0 [3 to 46]

5. Primary Outcome: Mean Difference in Change of Week 12 Value From Baseline of Participant-reported Total Symptom Interference Score From the MD Anderson Symptom Inventory (MDASI) Core Items
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: The ITT population included all randomized participants.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Atezolizumab Regimen | Atezolizumab Regimen + DPM
Number analyzed (Participants) | 25 | 24
Units on a scale
  Baseline: number analyzed (Participants) | 25 | 20
  Baseline | 3.33 [0.0 to 9.8] | 3.08 [0.0 to 9.5]
  Cycle 5 Day 1 (Week 12): number analyzed (Participants) | 15 | 15
  Cycle 5 Day 1 (Week 12) | 3.00 [0.0 to 9.0] | 2.33 [0.0 to 7.0]

ADVERSE EVENTS:
Time Frame: Up to approximately 16 months
Arm/Group | Atezolizumab Regimen | Atezolizumab Regimen + DPM
All-Cause Mortality (participants affected / at risk) | 6/25 | 2/24
Serious Adverse Events (participants affected / at risk) | 10/25 | 13/24
Other Adverse Events (participants affected / at risk) | 18/25 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab Regimen (N=25) | Atezolizumab Regimen + DPM (N=24)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab Regimen (N=25) | Atezolizumab Regimen + DPM (N=24)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 6 (8)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (3)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 3 (3)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (9)
Asthenia (General disorders) | 5 (5) | 3 (3)
Fatigue (General disorders) | 2 (2) | 7 (8)
Mucosal inflammation (General disorders) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 4 (4)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (3)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Proteinuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT05694013/Prot_SAP_000.pdf